CLINICAL TRIAL: NCT02628145
Title: Effects of a Resistance Training Program in Older Women With Sarcopenia
Acronym: RESTORE-ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Principal Investigator, Matthew J. Delmonico, PhD, MPH, Associate Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HU1415-168
Record Dates: First submitted 2015-12-01; First posted 2015-12-11 (Estimated); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2022-12

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; aging; resistance training; physical functioning
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resistance Training Intervention (Experimental): The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines follow American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Interventions: Behavioral: Resistance Training Intervention
- Active Control Group (Active Comparator): The CON group will meet three times weekly for approximately 12 weeks for light physical activity and stretching.
  Interventions: Behavioral: Active Control Group

INTERVENTIONS:
Behavioral: Resistance Training Intervention — The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is a NSCA certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations intensity are based on training phase. E.g., the first portion of 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and few unilateral and multi-joint light free weight exercise. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
  Arms: Resistance Training Intervention
Behavioral: Active Control Group — The CON group will meet three times weekly for approximately 12 weeks for light physical activity and stretching.
  Arms: Active Control Group

SUMMARY:
This is a randomized clinical trial with a control group that will test how periodized resistance training will impact measures of sarcopenia in older women who have been identified as presarcopenic or sarcopenic. The intervention will be approximately 12 weeks in duration with 24 total free-living older women. Outcome measures will be collected at baseline, 6 weeks and post-intervention.

DETAILED DESCRIPTION:
New sarcopenia (i.e. the age-related loss of muscle mass) guidelines established in 2014 recommend identifying older individuals for interventions who have low muscle strength and/or gait speed as these functional measures are associated with low muscle mass and subsequent negative health consequences such as increased mortality risk. Moreover, consensus guidelines indicate that more research, especially in older women, needs to be conducted to test the efficacy of periodized (i.e. planned variations in the program) resistance exercise training (RT) protocols in individuals who have been identified as sarcopenic or at risk of sarcopenia. Our interdisciplinary research group has conducted and published the results of several intervention studies in older adults and would like to expand this line of research to fill a critical gap in the current research. The broad objective of this research project is to help determine the efficacy of a periodized RT intervention strategy to treat sarcopenia or presarcopenia and its correlates among older women. The specific primary aim is to determine if there is significant effect of a RT program for improving physical functioning and muscle mass in older women. Exploratory aims are determine the impact of the RT intervention on other measures including bone density, lipoproteins, and other health indicators. The long-term goal of this project is to generate essential data for the submission of a more comprehensive NIH or private agency grant. The research design will be a randomized trial with a control group and methodology of this study will include 25 community-dwelling older women (age 65-84 years) for a 12-week repeated measures (baseline, 6 week, and post) randomized study with a six month observational follow-up. After baseline testing, participants will be randomized to either a RT intervention group (RTI) or to an active control (CON) group. The RT intervention will take place three times per week on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines follow American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults. The CON group will meet three times weekly for light physical activity and stretching. The relevance of this research is very significant as no studies to date have specifically examined RT in older women who have been identified as sarcopenic or presarcopenic using newly established guidelines. This study will accept all potential participants meeting inclusion criteria, regardless of ethnic, racial, or religious backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* Women, aged 65-84 years;
* Low lean mass and/or low physical functioning based on current guidelines;
* Currently (≥ 6 months) not engaged in a regular exercise program;
* Post-menopausal by self-report.

Exclusion Criteria:

* Failure to provide informed consent;
* Significant or suspected cognitive impairment;
* Severe hearing loss, speech disorder, language barrier or visual impairment;
* Progressive, degenerative neurologic disease;
* Terminal illness with life expectancy of < 12 months, as determined by a physician;
* Severe pulmonary disease, uncontrolled diabetes, blood pressure, or anemia;
* Medications not taken for > 3 weeks, lipid lowering medications for > 6 months;
* Major joint, vascular, abdominal, or thoracic surgery within six months;
* Significant cardiovascular disease or implanted pacemaker/defibrillator;
* Inability to safely engage in mild to moderate exercise with muscular exertion.

Ages: 65 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mattthew J Delmonico, PhD, Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Resistance Training Intervention | Active Control Group
Started | 13 | 12
Completed | 12 | 10
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Resistance Training Intervention | Active Control Group | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.8 (4.8) | 72.9 (4.6) | 72.3 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 12 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Muscle Mass Change: From Dual Energy X-ray Absorptiometry and Bioelectrical Impedance Analsysis - Appendicular Lean Mass (ALM in kg) Divided by Height (Meters-squared)
Description: Overall body composition was estimated using dual-energy x-ray absorptiometry (DXA) using fan-beam technology on a GE Lunar iDXA machine (GE, Waukesha, WI). Participants reported to testing in a fasted state (~12 hours) and wore surgical scrubs during the test. Standardized positioning procedures were followed and a licensed radiology technician performed all tests. Appendicular lean mass, total body fat mass, and percent fat were measured. Appendicular lean mass was considered the sum of non-bone lean mass in both arms and legs. Total body lean mass was defined as lean soft tissue mass plus total body bone mineral content.
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: kg/m2
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations intensity are based on the training phase. E.g., the first portion of the 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and a few unilateral and multi-joint light free weight exercises. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
kg/m2 | 0.09 (0.08) | 0.10 (0.09)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Other; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = -0.01

2. Secondary Outcome: Sarcopenia Status Change
Description: The multiple measurements will be aggregated to arrive at one reported value of change in the number of sarcopenic women using the International Working Group on Sarcopenia guidelines. Appendicular lean mass divided by height in meters squared <5.67 and gait speed of <1.0 meters per second indicates sarcopenia present. Change in status in 12 weeks indicates 1) stayed sarcopenic, 2) stayed non-sarcopenic, 3), became sarcopenic, or 4) became non-sarcopenic.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
Participants
  Stayed Sarcopenic | 7 | 5
  Stayed Non-Sarcopenic | 3 | 3
  Became Sarcopenic | 0 | 0
  Became Non-Sarcopenic | 2 | 2
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p = 0.88, Chi-squared

3. Secondary Outcome: Balance Ability: Single-leg Stand. Scored Yes or No
Description: Yes is a good outcome to be able to stand on one leg for 10 seconds. Categories for change in this in this ability are 1) Maintained Single Leg Stand Ability, 2) Maintained Single Leg Stand Inability, 3) Developed Single Leg Stand Ability, 4) Lost Single Leg Stand Ability.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations are based on the training phase. E.g., the first portion of the 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and a few unilateral and multi-joint light free weight exercises. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
Participants
  Maintained Single Leg Stand Ability | 5 | 4
  Maintained Single Leg Stand Inability | 3 | 4
  Developed Single Leg Stand Ability | 3 | 2
  Lost Single Leg Stand Ability. | 1 | 0
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p = 0.068, Fisher Exact

4. Secondary Outcome: Mobility Change: 8 Foot Timed up and go From a Seated Position Around a Cone Back to a Seated Position
Time Frame: 12 weeks
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
seconds | -0.48 (0.25) | -0.74 (0.27)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p = 0.48, Mixed Models Analysis

5. Secondary Outcome: Hip Bone Mineral Density: Measured by Dual Energy X-ray Absorptiometry
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: g/m2
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA-certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations intensity are based on the training phase. E.g., the first portion of the 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and a few unilateral and multi-joint light free weight exercises. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
g/m2 | -0.0005 (0.0197) | 0.0105 (0.0548)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p = 0.52, Mixed Models Analysis

6. Secondary Outcome: Physical Functioning Change: Normal Gait Speed Time From 400-meter Walk
Description: Change in timed 400-meter walk in seconds doing laps in a measured corridor at a pace that the participant can maintain.
Time Frame: 6 weeks, 12 weeks, and six month follow-up
Measure: Mean (Standard Error); unit: seconds
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations intensity is based on training phase. E.g., the first portion of the 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and a few unilateral and multi-joint light free weight exercises. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
seconds
  6 weeks | -14.28 (7.08) | -20.23 (8.07)
  12 weeks | -18.95 (8.53) | -20.89 (9.34)
  six month follow up | -14.61 (8.54) | -23.68 (9.36)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p > 0.05, Mixed Models Analysis

7. Secondary Outcome: Grip Strength Change: From Hand Grip Dynamometry in kg
Description: Handgrip strength was measured in both hands with the participant in a seated position using a handgrip dynamometer and standardized protocols (Jamar Hydraulic Dynamometer, J.A. Preston, Corp., Jackson, MS). Two trials per hand were completed and the highest score measured was used for sarcopenia classification.
Time Frame: 6 weeks, 12 weeks, and six month follow-up
Measure: Mean (Standard Error); unit: kg
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
kg
  6 weeks | 1.08 (0.90) | 1.45 (1.03)
  12 weeks | 1.67 (1.03) | 0.50 (1.26)
  six month follow up | 0.25 (0.95) | -0.10 (1.04)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p > 0.05, Mixed Models Analysis

8. Secondary Outcome: Muscle Strength Change: Leg Press One-repetition Maximum in kg
Description: All participants completed a familiarization with leg press machine one week prior to strength testing. Participants completed a set of 3-5 repetitions on the machine using a load determined by the participant to be comfortable, then a second set of 3-5 repetitions at an increased intensity, followed by 1-3 sets of progressively increasing intensity until the participant reached 80-90% of their maximal effort as rated on the Borg CR-10 scale. Maximal leg press strength was assessed using previously published methods on Cybex seated leg press machine (Cybex International Inc., Medway, MA). Participants completed a dynamic warm-up prior to strength testing. The leg press test required the participant to extend their knees from a starting position of ~90 degrees until the legs are fully extended, but not locked at the knees.
Time Frame: 6 weeks, 12 weeks, and six month follow-up
Population: Two participants from each group chose not to be retested.
Measure: Mean (Standard Error); unit: kg
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations intensity are based on training phase. E.g., the first portion of 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and few unilateral and multi-joint light free weight exercise. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
kg
  6 weeks | 13.35 (2.71) | 10.95 (2.96)
  12 weeks | 20.85 (3.41) | 17.93 (3.74)
  six month follow-up: number analyzed (Participants) | 10 | 8
  six month follow-up | 15.1 (2.97) | 12.50 (3.32)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p > 0.05, Mixed Models Analysis

9. Secondary Outcome: Chair Stand Time Change: Time to Complete Five Chair Rises From a Normal Chair
Time Frame: 6 weeks, 12 weeks, and six month follow-up
Population: Missing data or participants chose not to be retested.
Measure: Mean (Standard Error); unit: seconds
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
seconds
  6 weeks: number analyzed (Participants) | 12 | 9
  6 weeks | -0.95 (0.78) | -1.05 (0.90)
  12 weeks: number analyzed (Participants) | 11 | 10
  12 weeks | -1.56 (1.05) | -2.39 (1.10)
  six month follow-up | -1.13 (0.88) | -2.70 (1.00)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p > 0.05, Mixed Models Analysis

10. Secondary Outcome: Chair Stand Ability: Ability to Rise From a Chair One Time - Yes or No
Description: Chair stand ability: ability to rise from a chair one time - Yes or No, with "Yes" being a positive outcome. Two categories: 1) Able to Rise from a Chair and 2) Unable to Rise from a Chair
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
Participants
  Able to Rise from a Chair | 12 | 10
  Unable to Rise from a Chair | 0 | 0

11. Other Pre Specified Outcome: Body Mass Index Change: Weight in kg Divided by Height
Time Frame: 12 weeks
Population: Missing data point at week 12.
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
kg/m2 | 0.428 (0.423) | 0.007 (0.472)
Statistical Analysis 1: Comparison: Resistance Training Intervention vs Active Control Group; Test type: Superiority; p = 0.04, Mixed Models Analysis

12. Other Pre Specified Outcome: Body Mass, Baseline Only.
Description: Body mass in kg as measured from a balance-beam scale.
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
kg | 68.7 (15.5) | 61.8 (10.3)

13. Other Pre Specified Outcome: Height
Description: Height, measured in cm from a stadiometer
Time Frame: Baseline only
Measure: Mean (Standard Deviation); unit: cm
Groups:
- Resistance Training Intervention: The RT intervention will take place three times per week for approximately 12 weeks on non-consecutive days using 8-10 exercises for major muscle groups utilizing free weights and machines following American College of Sports Medicine and National Strength and Conditioning Association guidelines for RT in older adults.
  Resistance Training Intervention: The RTI group will participate in a periodized RT program on 3 non-consecutive days/week using NSCA and ACSM guidelines and will be designed by a team member who is an NSCA-certified strength and conditioning specialist. This program will consist of a full-body, nonlinear periodized program: a training method that has frequent variations in program variables. Intensity variations are based on the training phase. E.g., the first portion of 12-week cycle has more moderate and light days as participants adapt to the program. Weeks 1-4 will consist of primarily RT machine exercises and a few unilateral and multi-joint light free weight exercises. Weeks 5-8 will incorporate more free-weight exercises that are multi-joint. Weeks 9-12 will incorporate more complex multi-joint movements.
Arm/Group | Resistance Training Intervention | Active Control Group
Number analyzed (Participants) | 12 | 10
cm | 159.8 (5.9) | 159.7 (5.2)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Resistance Training Intervention | Active Control Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No